CLINICAL TRIAL: NCT04968028
Title: An Open-label Randomized Multi-centre Study to Evaluate Anterior Controllable Antedisplacement and Fusion Versus Posterior Laminoplasty in Patients With Cervical Ossification of the Posterior Longitudinal Ligament
Brief Title: Multi-centre Study to Evaluate ACAF Versus Laminoplasty in Treating Cervical Ossification of the Posterior Longitudinal Ligament
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Changhai Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tongji Hospital (Other); Peking University Shenzhen Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Xuanwu Hospital, Beijing (Other); Jining Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shanxi Bethune Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SL029
Record Dates: First submitted 2021-07-11; First posted 2021-07-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ossification of Posterior Longitudinal Ligament; Cervical Spondylosis With Myelopathy
Keywords: OPLL; Cervical Spondylotic Myelopathy; ACAF; Laminoplasty; Multicenter Study
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament | interventions — Gene Fusion; Laminoplasty

STUDY DESIGN:
Masking Description: In view of the obvious differences between the two surgery methods, this study was designed as an open-label trial. However, the results of X-ray, computed tomography (CT) and magnetic resonance imaging (MRI) will be independently reviewed by an independent radiographic review committee in a blind fashion in addition to the evaluation by site investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACAF (Experimental): Participants underwent anterior decompression of Anterior Controllable Antedisplacement and Fusion
  Interventions: Procedure: ACAF
- Laminoplasty (Experimental): Participants underwent posterior decompression of Laminoplasty
  Interventions: Procedure: Laminoplasty

INTERVENTIONS:
Procedure: ACAF — (1)A standard right-side Smith-Robinson approach is performed. (2) The involved disc tissues are removed. The posterior longitudinal ligament is cut down at the levels cephalic and caudal to OPLL. (3) The anterior portion of the middle vertebral bodies is removed according to the thickness of ossification. Suitable cages are placed into each intervertebral space. (4) On the left side of the vertebra, a 2-mm-wide groove is created at the medial border of the transverse foramina. After that, an curved plated is fixed with screws. (5) On the right side of the vertebrae, a similar groove was also created. (6) Finally, tightening the screws to achieve a gradual evaluation of the vertebrae with OPLL.
  Other Names: Anterior Controllable Antedisplacement and Fusion
  Arms: ACAF
Procedure: Laminoplasty — (1) In the prone position, the skin and nuchal ligament were cut through the posterior median incision, and the paravertebral muscles were stripped layer by layer to expose the bilateral vertebral lamina, lateral mass and articular process.（2) Part of spinous process were removed with bone biting forceps. The side with more severe symptoms was selected as the open side, bone groove was performed at 2-3 mm of the medial edge of bilateral facet joints with the medial cortex was reserved at the shaft side.（3) Slowly lift the lamina and maintained.（4)Determining the opening width of each segment by trial, and selecting the appropriate size Arch miniplate, and fixed with screws.
  Arms: Laminoplasty

SUMMARY:
The purpose of this study is to compare the efficacy, safety and imaging outcomes between Anterior Controllable Antedisplacement and Fusion (ACAF) and Laminoplasty in the treatment of severe ossification of cervical posterior longitudinal ligament.

DETAILED DESCRIPTION:
This is a national, multicenter, prospective, randomized controlled trial to compare the safety and efficacy of ACAF and posterior laminoplasty in the treatment of severe ossification of cervical posterior longitudinal ligament. In this study, 164 adult patients aged 18-70 with severe copll were randomly assigned to the experimental group (using ACAF) and the control group (using lamp) according to the ratio of 1:1. The patients were followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age is 18-70 years old, regardless of gender;
2. The patient was diagnosed as severe ossification of the posterior longitudinal ligament (X-ray or CT showed ossification of the posterior longitudinal ligament); The imaging findings showed occupied ratio ≥ 60% or involved three or more segments;
3. Symptoms of spinal cord and nerve root compression, or accompanied by spinal cord compression symptoms such as dysfunction of urination and defecation, conservative treatment was ineffective or aggravated gradually;
4. The participant (or his legal guardian) can sign the informed consent.

Exclusion Criteria:

1. Congenital malformations (including but not limited to occipitocervical malformations, congenital cervical fusion, cervical related neurovascular malformations), ossification of cervical ligamentum flavum, cervical trauma, cervical cancer, cervical tuberculosis and other inflammatory diseases;
2. Patients with other spinal diseases such as thoracolumbar vertebrae that affect clinical symptoms; Patients with motor neuron diseases such as amyotrophic lateral sclerosis and other nervous system diseases;
3. The symptoms were aggravated due to recent trauma;
4. Patients who participated in other clinical trials in recent 3 months;
5. The participant (or his legal guardian) with mental illness and cognitive impairment can not give full informed consent;
6. Those who are in poor health and can not tolerate surgery; The patients were not suitable for surgical treatment after preoperative examination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
C-JOA Recovery Rate | Time point of outcome: 3 months post-operative follow-up visits
  (postoperative JOA score at 3 months follow-up - preoperative JOA score)/(17 - preoperative JOA score)* 100%
C-JOA Recovery Rate | Time point of outcome: 6 months post-operative follow-up visits
  (postoperative JOA score at 6 months follow-up - preoperative JOA score)/(17 - preoperative JOA score)* 100%
C-JOA Recovery Rate | Time point of outcome: 12 months post-operative follow-up visits
  (postoperative JOA score at 12 months follow-up - preoperative JOA score)/(17 - preoperative JOA score)* 100%
C-JOA Recovery Rate | Time point of outcome: 24 months post-operative follow-up visits
  (postoperative JOA score at 24 months follow-up - preoperative JOA score)/(17 - preoperative JOA score)* 100%

SECONDARY OUTCOMES:
Japanese Orthopaedic Association Scores | 28 days before operation and 3, 6, 12, 24 months post-operative follow-up visits
  Filling in the Japanese Orthopaedic Association Scores scale. This scale involves four aspects: upper limb motor function (range, 0 to 4 points), lower limb motor function (range, 0 to 4 points), sensory function (range, 0 to 6 points), and bladder function (range, 0 to 3 points). The total C-JOA score ranged from 0 (worst) to 17 (normal condition).
Visual Analogue Scale | 28 days before operation and 3, 6, 12, 24 months post-operative follow-up visits
  Filling in the Visual Analogue Scale pain score that range, 0 [no pain] to 10 [most severe].
Neck Disability Index | 28 days before operation and 3, 6, 12, 24 months post-operative follow-up visits
  Filling in the 10-item Neck Disability Index scale that totally range 0 to 50 points, the highest index the worst.
Nurick-Score | 28 days before operation and 3, 6, 12, 24 months post-operative follow-up visits
  Filling in the 6-level Nurick disability grade scale that range 0 [mild] to 5 [severe].

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Shi, Doctor, Study Chair — Shanghai Changzheng Hospital; Dan Han, Master, Study Director — Shanghai Changzheng Hospital; Yu Chen, Doctor, Principal Investigator — Shanghai Changzheng Hospital
Locations (12):
- China (12):
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjaing
  - Xuanwu Hospital Capital Medical University, Beijing, Pekin
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital, Air Force Medical University, Xi’an, Shanxi

REFERENCES:
- [Background] Chen Y, Sun J, Yuan X, Guo Y, Yang H, Chen D, Shi J. Comparison of Anterior Controllable Antedisplacement and Fusion With Posterior Laminoplasty in the Treatment of Multilevel Cervical Ossification of the Posterior Longitudinal Ligament: A Prospective, Randomized, and Control Study With at Least 1-Year Follow Up. Spine (Phila Pa 1976). 2020 Aug 15;45(16):1091-1101. doi: 10.1097/BRS.0000000000003462. PMID 32097261
- [Background] Sun K, Wang S, Huan L, Sun J, Xu X, Sun X, Shi J, Guo Y. Analysis of the spinal cord angle for severe cervical ossification of the posterior longitudinal ligament: comparison between anterior controllable antedisplacement and fusion (ACAF) and posterior laminectomy. Eur Spine J. 2020 May;29(5):1001-1012. doi: 10.1007/s00586-019-06216-6. Epub 2019 Dec 3. PMID 31797138
- [Derived] Chen Y, Sun J, Han D, Yuan X, Wang Y, Guo Y, Zhong X, Shi J. An open-label randomized multi-Centre study to evaluate anterior controllable Antedisplacement and fusion versus posterior Laminoplasty in patients with cervical ossification of the posterior longitudinal ligament: study design and analysis plan (STAR). BMC Musculoskelet Disord. 2021 Sep 8;22(1):765. doi: 10.1186/s12891-021-04645-3. PMID 34496821